CLINICAL TRIAL: NCT04526158
Title: Testing Two Scalable, Veteran-centric Mindfulness-based Interventions for Chronic Musculoskeletal Pain: A Pragmatic, Multisite Trial
Brief Title: Learning to Apply Mindfulness to Pain
Acronym: LAMP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Principal Investigator, Diana J. Burgess, Principal Investigator, Minneapolis Veterans Affairs Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: #NH170001
Record Dates: First submitted 2020-07-09; First posted 2020-08-25 (Actual); Results first posted 2024-11-05 (Actual); Last update posted 2024-11-05 (Actual); Status verified 2024-10

CONDITIONS: Chronic Pain
Keywords: Mindfulness; Veteran; Chronic pain
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Intervention Model Description: Three arm parallel assignment design
Masking Description: The randomization list will be concealed from the research team within the tracking portal, so team members will not know the next study assignment. Permuted blocks will be used to aid in the concealment of treatment assignment while ensuring balance in treatment arms across time.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Mobile+Group LAMP Mindfulness-Based Intervention (Experimental): 8 weekly, synchronous interactive online group sessions; access to mobile app and a study website, with an accompanying workbook.
  Interventions: Behavioral: Mobile+Group LAMP Mindfulness-Based Intervention
- Mobile LAMP Mindfulness-Based Intervention (Experimental): 8 weekly asynchronous sessions, delivered on mobile app and study website, with an accompanying workbook; 3 engagement calls at the middle, beginning and end of the program.
  Interventions: Behavioral: Mobile LAMP Mindfulness-Based Intervention
- Usual Care (No Intervention): Engagement in usual care for 12 months as participants normally would. After the entire follow-up period is complete (12 months), participants in the usual care arm are given access to the Mobile LAMP materials MBI training on the app and study website, and the accompanying workbook.

INTERVENTIONS:
Behavioral: Mobile+Group LAMP Mindfulness-Based Intervention — The Mobile+Group LAMP Mindfulness-Based Intervention (MBI) condition consists of eight 90-minute weekly group sessions, delivered via secure video-conferencing. The first session is preceded by a 90-minute technical session introducing the video-conference system and other logistics. The program consists of educational and instructional videos presented by a trained mindfulness instructor interspersed with workbook reflections and group discussions, and daily practice exercises that participants do on their own. A trained facilitator (who is not required to be an expert in mindfulness) leads the group. Participants also have access to a mobile app and a study website, with the same educational and instructional videos that are presented in the group sessions, and the accompanying workbook.
  Other Names: Mobile+Group LAMP
  Arms: Mobile+Group LAMP Mindfulness-Based Intervention
Behavioral: Mobile LAMP Mindfulness-Based Intervention — The Mobile LAMP MBI consists of 8 self-paced, 30- to 60-minute weekly sessions, delivered on a mobile app and available on the study website, with an accompanying workbook. The program consists of educational and instructional videos presented by a trained mindfulness instructor, with workbook reflections and daily practice exercises that participants do on their own (the same content used in Mobile+Group LAMP). Participants also participate in 3 engagement phone calls with a facilitator. The 1st call (45-60 minutes), held at the beginning of the program, includes technical and logistical information on engaging with mobile app, website, and workbook; and discussion of goals, challenges and plans for practice. The 2nd (middle of program) and 3rd call (end of program) are 25-45 minutes long and address technical/logistical issues and discussion of goals, progress, plans for practice and strategies to address challenges.
  Other Names: Mobile LAMP
  Arms: Mobile LAMP Mindfulness-Based Intervention

SUMMARY:
The long-term goal of this two-phase project is to reduce chronic pain and co-morbid conditions among Veterans, through scalable, non-pharmacologic evidence-based strategies that are "Veteran-Centric," designed to optimize engagement, adherence and sustainability, and are deliverable to large numbers of Veterans.

DETAILED DESCRIPTION:
The investigators will conduct a 3-site 3-arm pragmatic clinical trial (N = 750) to test effectiveness of 2 Mindfulness-Based Interventions (MBIs), Mobile+Group LAMP and Mobile LAMP, compared to usual practice. Effectiveness will be assessed by pain functioning over the 12-month follow-up period using the Brief Pain Inventory (BPI) interference score. The investigators will test the following primary hypotheses: (1) Mobile LAMP will be more effective at improving chronic pain (as measured by change in the BPI interference score over the 12-month follow-up period) compared to usual practice, (2) Mobile+Group LAMP will be more effective at improving chronic pain (as measured by BPI interference score over the 12-month follow-up period) compared to usual practice, and (3) Mobile+Group LAMP will be more effective at improving chronic pain (as measured by BPI interference change over the 12-month follow-up period) compared to Mobile LAMP without the group component. The investigators will test the following secondary hypotheses: (1) Comparison of intervention group with secondary outcomes listed below, and (2) primary and secondary hypotheses comparisons will be confirmed in gender-specific strata. The primary outcome will be measured as change in BPI interference score over the 12-month follow-up period. Secondary outcomes will include patient-reported measures related to pain, comorbid mental health conditions and function, expected mediators of treatment effects, patient satisfaction, and adverse effects and measures captured in electronic health records. These outcomes will be assessed at 10 weeks, 6 months and 12 months. Implementation data will be collected and described, using the guided Reach, Effectiveness, Adoption, Implementation, and Maintenance (RE-AIM) framework.

ELIGIBILITY:
Inclusion Criteria:

* Must have qualifying pain diagnoses on at least 2 occasions, at least 90 days apart, within the same pain category, during the previous 2 years
* Must report having a pain duration of ≥ 6 months (pain chronicity threshold), and a pain severity score of ≥ 4 on the 0-10 Numeric Rating Scale (pain severity threshold).
* Must have access to a smart phone that meets the requirement of the mobile app software
* Must be willing and able to download the mobile app on their phone
* Must have wireless or cellular internet access on a daily basis
* Must be willing to meet via video conference on the dates and at the time when Mobile+Group LAMP sessions are held, and attend all sessions of the arm to which they are randomized.

Exclusion Criteria:

* new diagnosis of schizophrenia, bipolar disorder, major depressive disorder, or other psychosis within the past 18 months; or current active psychotic symptoms, suicidality, severe depression, manic episode, and/or poorly controlled bipolar disorder (as assessed by a medical chart review)
* currently enrolled in a research study for pain
* currently enrolled in mindfulness-based stress reduction (MBSR)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 811 (Actual)
Dates: Start 2020-11-02 (Actual); Primary Completion 2023-08-30 (Actual); Study Completion 2023-12-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Minnesota Veteran Administration Health Care System, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Burgess DJ, Evans R, Allen KD, Bangerter A, Bronfort G, Cross LJ, Ferguson JE, Haley A, Hagel Campbell EM, Mahaffey MR, Matthias MS, Meis LA, Polusny MA, Serpa JG, Taylor SL, Taylor BC. Learning to Apply Mindfulness to Pain (LAMP): Design for a Pragmatic Clinical Trial of Two Mindfulness-Based Interventions for Chronic Pain. Pain Med. 2020 Dec 12;21(Suppl 2):S29-S36. doi: 10.1093/pm/pnaa337. PMID 33313730
- [Background] Burgess DJ, Calvert C, Hagel Campbell EM, Allen KD, Bangerter A, Behrens K, Branson M, Bronfort G, Cross LJS, Evans R, Ferguson JE, Friedman JK, Haley AC, Leininger B, Mahaffey M, Matthias MS, Meis LA, Polusny MA, Serpa JG, Taylor SL, Taylor BC. Telehealth Mindfulness-Based Interventions for Chronic Pain: The LAMP Randomized Clinical Trial. JAMA Intern Med. 2024 Oct 1;184(10):1163-1173. doi: 10.1001/jamainternmed.2024.3940. PMID 39158851
- [Derived] Burgess DJ, Calvert C, Bangerter A, Branson M, Cross LJS, Evans R, Ferguson JE, Friedman JK, Hagel Campbell EM, Haley AC, Hennessy S, Kraft C, Mahaffey M, Matthias MS, Meis LA, Serpa JG, Taylor SL, Taylor BC. Do mindfulness interventions cause harm? Findings from the Learning to Apply Mindfulness to Pain (LAMP) Pragmatic Clinical Trial. Pain Med. 2024 Nov 1;25(Supplement_1):S68-S76. doi: 10.1093/pm/pnae056. PMID 39514882
- [Derived] Ferguson JE, Hagel Campbell E, Bangerter A, Cross LJS, Allen KD, Behrens K, Branson M, Calvert C, Friedman JK, Hennessy S, Meis LA, Taylor BC, Burgess DJ. Email recruitment for chronic pain clinical trials: results from the LAMP trial. Trials. 2024 Jul 19;25(1):491. doi: 10.1186/s13063-024-08301-8. PMID 39030622
- [Derived] Burgess DJ, Hagel Campbell EM, Branson M, Calvert C, Evans R, Allen KD, Bangerter A, Cross LJS, Driscoll MA, Hennessy S, Ferguson JE, Friedman JK, Matthias MS, Meis LA, Polusny MA, Taylor SL, Taylor BC. Exploring Gender Differences in Veterans in a Secondary Analysis of a Randomized Controlled Trial of Mindfulness for Chronic Pain. Womens Health Rep (New Rochelle). 2024 Feb 12;5(1):82-92. doi: 10.1089/whr.2023.0086. eCollection 2024. PMID 38404673

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Mobile+Group LAMP Mindfulness-Based Intervention | Mobile LAMP Mindfulness-Based Intervention | Usual Care
Started | 270 | 271 | 270
Completed | 225 | 225 | 244
Not Completed | 45 | 46 | 26

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Mobile+Group LAMP Mindfulness-Based Intervention | Mobile LAMP Mindfulness-Based Intervention | Usual Care | Total
Number analyzed (Participants) | 270 | 271 | 270 | 811
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.2 (13.3) | 55.7 (13.0) | 55.0 (12.2) | 54.6 (12.9)
Sex: Female, Male [Count of Participants; unit: Participants] — Operationalized as gender; woman, man
  Participants
    Female | 133 | 128 | 126 | 387
    Male | 137 | 143 | 144 | 424
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 15 | 16 | 20 | 51
  Not Hispanic or Latino | 255 | 254 | 250 | 759
  Unknown or Not Reported | 0 | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 2 | 6 | 10
  Asian | 1 | 3 | 2 | 6
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 0 | 1
  Black or African American | 73 | 68 | 67 | 208
  White | 182 | 184 | 180 | 546
  More than one race | 9 | 14 | 13 | 36
  Unknown or Not Reported | 2 | 0 | 2 | 4
Region of Enrollment [Number; unit: participants]
  United States | 270 | 271 | 270 | 811

OUTCOME MEASURES:

1. Primary Outcome: Change in the Brief Pain Inventory (BPI) Interference Score From Baseline, Over the 12-month Follow-up Period.
Description: Change in the Brief Pain Inventory (BPI) interference score. Minimum value: 0. Maximum value: 10. Higher scores indicate worse functioning.
  Change in the outcome measure operationalized as the weighted average of all of the time points during follow-up, adjusting for the baseline value prior to randomization.
Time Frame: Weighted average over 10 weeks, 6 months, and 12 months.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Mobile+Group LAMP Mindfulness-Based Intervention | Mobile LAMP Mindfulness-Based Intervention | Usual Care
Number analyzed (Participants) | 270 | 271 | 270
score on a scale | 4.8 (0.1) | 4.5 (0.1) | 5.2 (0.1)
Statistical Analysis 1: Comparison: Mobile+Group LAMP Mindfulness-Based Intervention vs Mobile LAMP Mindfulness-Based Intervention; Test type: Superiority; p = 0.031, Mixed Models Analysis — significance threshold = 0.0167 due to multiple comparisons; Linear mixed model adjusted for baseline values of BPI interference, Pain Self-Efficacy, and design factors; Mean Difference (Final Values) = 0.3, 95% CI 2-sided [0.0 to 0.6] — estimates were generated from multiple imputed data
Statistical Analysis 2: Comparison: Mobile+Group LAMP Mindfulness-Based Intervention vs Usual Care; Test type: Superiority; p = 0.002, Mixed Models Analysis — significance threshold = 0.0167 due to multiple comparisons; Linear mixed model adjusted for baseline values of BPI interference, Pain Self-Efficacy, and design factors; Mean Difference (Final Values) = -0.4, 95% CI 2-sided [-0.7 to -0.2] — estimates were generated from multiple imputed data
Statistical Analysis 3: Comparison: Mobile LAMP Mindfulness-Based Intervention vs Usual Care; Test type: Superiority; p < 0.001, Mixed Models Analysis — significance threshold = 0.0167 due to multiple comparisons; Linear mixed model adjusted for baseline values of BPI interference, Pain Self-Efficacy, and design factors; Mean Difference (Final Values) = -0.7, 95% CI 2-sided [-1.0 to -0.4] — estimates were generated from multiple imputed data

2. Secondary Outcome: Change in the Brief Pain Inventory (BPI) Intensity Score From Baseline, Over the 12-month Follow-up Period.
Description: Brief Pain Inventory (BPI) intensity score. Minimum value: 0. Maximum value: 10. Higher scores indicate more severe pain. Change in the outcome measure operationalized as the weighted average of all of the time points during follow-up, adjusting for the baseline value prior to randomization.
Time Frame: Weighted average over 10 weeks, 6 months, and 12 months.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Mobile+Group LAMP Mindfulness-Based Intervention | Mobile LAMP Mindfulness-Based Intervention | Usual Care
Number analyzed (Participants) | 270 | 271 | 270
score on a scale | 4.7 (0.1) | 4.6 (0.1) | 5.1 (0.1)
Statistical Analysis 1: Comparison: Mobile+Group LAMP Mindfulness-Based Intervention vs Mobile LAMP Mindfulness-Based Intervention; Test type: Superiority; p = 0.736, Mixed Models Analysis; Linear mixed model adjusted for baseline values of BPI intensity, Pain Self-Efficacy, and design factors; Mean Difference (Final Values) = 0.0, 95% CI 2-sided [-0.2 to 0.3] — estimates were generated from multiple imputed data
Statistical Analysis 2: Comparison: Mobile+Group LAMP Mindfulness-Based Intervention vs Usual Care; Test type: Superiority; p < 0.001, Mixed Models Analysis; Linear mixed model adjusted for baseline values of BPI intensity, Pain Self-Efficacy, and design factors; Mean Difference (Final Values) = -0.4, 95% CI 2-sided [-0.6 to -0.2] — estimates were generated from multiple imputed data
Statistical Analysis 3: Comparison: Mobile LAMP Mindfulness-Based Intervention vs Usual Care; Test type: Superiority; p < 0.001, Mixed Models Analysis; Linear mixed model adjusted for baseline values of BPI intensity, Pain Self-Efficacy, and design factors; Mean Difference (Final Values) = -0.4, 95% CI 2-sided [-0.7 to -0.2] — estimates were generated from multiple imputed data

3. Secondary Outcome: Change in Physical Functioning Over the 12-month Follow-up Period Assessed by Mean Score on the Patient-Reported Outcomes Measurement Information System (PROMIS)-29 Profile v.2.0 Measure of Physical Function
Description: Patient-Reported Outcomes Measurement Information System (PROMIS)-29 Profile v.2.0 measure of physical function. Minimum value: 4. Maximum value: 20. Lower scores indicate worse physical functioning. Change in the outcome measure operationalized as the weighted average of all of the time points during follow-up, adjusting for the baseline value prior to randomization.
Time Frame: Weighted average over 10 weeks, 6 months, and 12 months.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Mobile+Group LAMP Mindfulness-Based Intervention | Mobile LAMP Mindfulness-Based Intervention | Usual Care
Number analyzed (Participants) | 270 | 271 | 270
score on a scale | 13.3 (0.1) | 13.3 (0.1) | 12.7 (0.1)
Statistical Analysis 1: Comparison: Mobile+Group LAMP Mindfulness-Based Intervention vs Mobile LAMP Mindfulness-Based Intervention; Test type: Superiority; p = 0.829, Mixed Models Analysis; Linear mixed model adjusted for baseline values of PROMIS Physical function, Pain Self-Efficacy, and design factors; Mean Difference (Final Values) = 0.0, 95% CI 2-sided [-0.4 to 0.4] — estimates were generated from multiple imputed data
Statistical Analysis 2: Comparison: Mobile+Group LAMP Mindfulness-Based Intervention vs Usual Care; Test type: Superiority; p = 0.005, Mixed Models Analysis; Linear mixed model adjusted for baseline values of PROMIS Physical function, Pain Self-Efficacy, and design factors; Mean Difference (Final Values) = 0.5, 95% CI 2-sided [0.2 to 0.9] — estimates were generated from multiple imputed data
Statistical Analysis 3: Comparison: Mobile LAMP Mindfulness-Based Intervention vs Usual Care; Test type: Superiority; p = 0.004, Mixed Models Analysis; Linear mixed model adjusted for baseline values of PROMIS Physical function, Pain Self-Efficacy, and design factors; Mean Difference (Final Values) = 0.6, 95% CI 2-sided [0.2 to 1.0] — estimates were generated from multiple imputed data

4. Secondary Outcome: Change in Anxiety Over the 12-month Follow-up Period Assessed by Mean Score on the Patient-Reported Outcomes Measurement Information System (PROMIS)-29 Profile v.2.0 Measure of Anxiety
Description: Patient-Reported Outcomes Measurement Information System (PROMIS)-29 Profile v.2.0 measure of anxiety. Minimum value: 4. Maximum value: 20. Higher scores indicate worse anxiety. Change in the outcome measure operationalized as the weighted average of all of the time points during follow-up, adjusting for the baseline value prior to randomization.
Time Frame: Weighted average over 10 weeks, 6 months, and 12 months.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Mobile+Group LAMP Mindfulness-Based Intervention | Mobile LAMP Mindfulness-Based Intervention | Usual Care
Number analyzed (Participants) | 270 | 271 | 270
score on a scale | 9.2 (0.1) | 8.8 (0.2) | 9.4 (0.1)
Statistical Analysis 1: Comparison: Mobile+Group LAMP Mindfulness-Based Intervention vs Mobile LAMP Mindfulness-Based Intervention; Test type: Superiority; p = 0.079, Mixed Models Analysis; Linear mixed model adjusted for baseline values of PROMIS Anxiety, Pain Self-Efficacy, and design factors; Mean Difference (Final Values) = 0.4, 95% CI 2-sided [0.0 to 0.8] — estimates were generated from multiple imputed data
Statistical Analysis 2: Comparison: Mobile+Group LAMP Mindfulness-Based Intervention vs Usual Care; Test type: Superiority; p = 0.296, Mixed Models Analysis; Linear mixed model adjusted for baseline values of PROMIS Anxiety, Pain Self-Efficacy, and design factors; Mean Difference (Final Values) = -0.2, 95% CI 2-sided [-0.6 to 0.2] — estimates were generated from multiple imputed data
Statistical Analysis 3: Comparison: Mobile LAMP Mindfulness-Based Intervention vs Usual Care; Test type: Superiority; p = 0.005, Mixed Models Analysis; Linear mixed model adjusted for baseline values of PROMIS Anxiety, Pain Self-Efficacy, and design factors; Mean Difference (Final Values) = -0.6, 95% CI 2-sided [-1.0 to -0.2] — estimates were generated from multiple imputed data

5. Secondary Outcome: Change in Fatigue Over the 12-month Follow-up Period Assessed by Mean Score on the Patient-Reported Outcomes Measurement Information System (PROMIS)-29 Profile v.2.0 Measure of Fatigue
Description: Patient-Reported Outcomes Measurement Information System (PROMIS)-29 Profile v.2.0 measure of fatigue. Minimum value: 4. Maximum value: 20. Higher scores indicate worse fatigue. Change in the outcome measure operationalized as the weighted average of all of the time points during follow-up, adjusting for the baseline value prior to randomization.
Time Frame: Weighted average over 10 weeks, 6 months, and 12 months.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Mobile+Group LAMP Mindfulness-Based Intervention | Mobile LAMP Mindfulness-Based Intervention | Usual Care
Number analyzed (Participants) | 270 | 271 | 270
score on a scale | 12.9 (0.2) | 12.7 (0.2) | 13.5 (0.2)
Statistical Analysis 1: Comparison: Mobile+Group LAMP Mindfulness-Based Intervention vs Mobile LAMP Mindfulness-Based Intervention; Test type: Superiority; p = 0.464, Mixed Models Analysis; Linear mixed model adjusted for baseline values of PROMIS fatigue, Pain Self-Efficacy, and design factors; Mean Difference (Final Values) = 0.2, 95% CI 2-sided [-0.3 to 0.7] — estimates were generated from multiple imputed data
Statistical Analysis 2: Comparison: Mobile+Group LAMP Mindfulness-Based Intervention vs Usual Care; Test type: Superiority; p = 0.019, Mixed Models Analysis; Linear mixed model adjusted for baseline values of PROMIS fatigue, Pain Self-Efficacy, and design factors; Mean Difference (Final Values) = -0.6, 95% CI 2-sided [-1.1 to -0.1] — estimates were generated from multiple imputed data
Statistical Analysis 3: Comparison: Mobile LAMP Mindfulness-Based Intervention vs Usual Care; Test type: Superiority; p = 0.002, Mixed Models Analysis; Linear mixed model adjusted for baseline values of PROMIS fatigue, Pain Self-Efficacy, and design factors; Mean Difference (Final Values) = -0.8, 95% CI 2-sided [-1.3 to -0.3] — estimates were generated from multiple imputed data

6. Secondary Outcome: Change in Sleep Disturbance Over the 12-month Follow-up Period Assessed by Mean Score on the Patient-Reported Outcomes Measurement Information System (PROMIS)-29 Profile v.2.0 Measure of Sleep Disturbance
Description: Patient-Reported Outcomes Measurement Information System (PROMIS)-29 Profile v.2.0 measure of sleep disturbance. Minimum value: 4. Maximum value: 20. Higher scores indicate worse sleep disturbance. Change in the outcome measure operationalized as the weighted average of all of the time points during follow-up, adjusting for the baseline value prior to randomization.
Time Frame: Weighted average over 10 weeks, 6 months, and 12 months.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Mobile+Group LAMP Mindfulness-Based Intervention | Mobile LAMP Mindfulness-Based Intervention | Usual Care
Number analyzed (Participants) | 270 | 271 | 270
score on a scale | 13.3 (0.2) | 13.3 (0.2) | 13.9 (0.2)
Statistical Analysis 1: Comparison: Mobile+Group LAMP Mindfulness-Based Intervention vs Mobile LAMP Mindfulness-Based Intervention; Test type: Superiority; p = 0.889, Mixed Models Analysis; Linear mixed model adjusted for baseline values of PROMIS sleep disturbance, Pain Self-Efficacy, and design factors; Mean Difference (Final Values) = 0.0, 95% CI 2-sided [-0.5 to 0.4] — estimates were generated from multiple imputed data
Statistical Analysis 2: Comparison: Mobile+Group LAMP Mindfulness-Based Intervention vs Usual Care; Test type: Superiority; p = 0.004, Mixed Models Analysis; Linear mixed model adjusted for baseline values of PROMIS sleep disturbance, Pain Self-Efficacy, and design factors; Mean Difference (Final Values) = -0.7, 95% CI 2-sided [-1.1 to -0.2] — estimates were generated from multiple imputed data
Statistical Analysis 3: Comparison: Mobile LAMP Mindfulness-Based Intervention vs Usual Care; Test type: Superiority; p = 0.006, Mixed Models Analysis; Linear mixed model adjusted for baseline values of PROMIS sleep disturbance, Pain Self-Efficacy, and design factors; Mean Difference (Final Values) = -0.6, 95% CI 2-sided [-1.1 to -0.2] — estimates were generated from multiple imputed data

7. Secondary Outcome: Change in Participation in Social Roles and Activities Over the 12-month Follow-up Period Assessed by Mean Score on the PROMIS-29 Profile v.2.0 Measure of Participation in Social Roles and Activities
Description: PROMIS-29 Profile v.2.0 measure of participation in social roles and activities. Minimum value: 4. Maximum value: 20. Lower scores indicate greater participation in social roles and activities. Change in the outcome measure operationalized as the weighted average of all of the time points during follow-up, adjusting for the baseline value prior to randomization.
Time Frame: Weighted average over 10 weeks, 6 months, and 12 months.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Mobile+Group LAMP Mindfulness-Based Intervention | Mobile LAMP Mindfulness-Based Intervention | Usual Care
Number analyzed (Participants) | 270 | 271 | 270
score on a scale | 12.0 (0.2) | 11.9 (0.2) | 11.0 (0.1)
Statistical Analysis 1: Comparison: Mobile+Group LAMP Mindfulness-Based Intervention vs Mobile LAMP Mindfulness-Based Intervention; Test type: Superiority; p = 0.76, Mixed Models Analysis; Linear mixed model adjusted for baseline values of PROMIS social roles and activities, Pain Self-Efficacy, and design factors; Mean Difference (Final Values) = 0.1, 95% CI 2-sided [-0.4 to 0.5] — estimates were generated from multiple imputed data
Statistical Analysis 2: Comparison: Mobile+Group LAMP Mindfulness-Based Intervention vs Usual Care; Test type: Superiority; p < 0.001, Mixed Models Analysis; [statistical method as in outcome 7, analysis 1]; Mean Difference (Final Values) = 1.0, 95% CI 2-sided [0.6 to 1.4] — estimates were generated from multiple imputed data
Statistical Analysis 3: Comparison: Mobile LAMP Mindfulness-Based Intervention vs Usual Care; Test type: Superiority; p < 0.001, Mixed Models Analysis; [statistical method as in outcome 7, analysis 1]; Mean Difference (Final Values) = 0.9, 95% CI 2-sided [0.5 to 1.3] — estimates were generated from multiple imputed data

8. Secondary Outcome: Change in Depression Over the 12-month Follow-up Period Assessed by Score on the Eight-item Patient Health Questionnaire Depression Scale (PHQ8)
Description: Patient Health Questionnaire depression scale (PHQ8). Minimum value: 0. Maximum value: 24. Higher scores indicate greater depression. Change in the outcome measure operationalized as the weighted average of all of the time points during follow-up, adjusting for the baseline value prior to randomization.
Time Frame: Weighted average over 10 weeks, 6 months, and 12 months.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Mobile+Group LAMP Mindfulness-Based Intervention | Mobile LAMP Mindfulness-Based Intervention | Usual Care
Number analyzed (Participants) | 270 | 271 | 270
score on a scale | 8.2 (0.2) | 8.2 (0.2) | 9.1 (0.2)
Statistical Analysis 1: Comparison: Mobile+Group LAMP Mindfulness-Based Intervention vs Mobile LAMP Mindfulness-Based Intervention; Test type: Superiority; p = 0.89, Mixed Models Analysis; Linear mixed model adjusted for baseline values of PHQ8, Pain Self-Efficacy, and design factors; Mean Difference (Final Values) = 0.0, 95% CI 2-sided [-0.7 to 0.6] — estimates were generated from multiple imputed data
Statistical Analysis 2: Comparison: Mobile+Group LAMP Mindfulness-Based Intervention vs Usual Care; Test type: Superiority; p = 0.003, Mixed Models Analysis; Linear mixed model adjusted for baseline values of PHQ8, Pain Self-Efficacy, and design factors; Mean Difference (Final Values) = -0.9, 95% CI 2-sided [-1.5 to -0.3] — estimates were generated from multiple imputed data
Statistical Analysis 3: Comparison: Mobile LAMP Mindfulness-Based Intervention vs Usual Care; Test type: Superiority; p = 0.007, Mixed Models Analysis; Linear mixed model adjusted for baseline values of PHQ8, Pain Self-Efficacy, and design factors; Mean Difference (Final Values) = -0.9, 95% CI 2-sided [-1.5 to -0.2] — estimates were generated from multiple imputed data

9. Secondary Outcome: Change in Post Traumatic Stress Disorder (PTSD), Over the 12-month Follow-up Period, Assessed by Participants' Scores on the Post Traumatic Stress Disorder Checklist for Diagnostic and Statistical Manual of Mental Disorders - 5 (PCL-5)
Description: Post Traumatic Stress Disorder Checklist for Diagnostic and Statistical Manual of Mental Disorders - 5 (PCL-5). Minimum value: 0. Maximum value: 80. Higher scores indicate greater PTSD. Change in the outcome measure operationalized as the weighted average of all of the time points during follow-up, adjusting for the baseline value prior to randomization.
Time Frame: Weighted average over 10 weeks, 6 months, and 12 months.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Mobile+Group LAMP Mindfulness-Based Intervention | Mobile LAMP Mindfulness-Based Intervention | Usual Care
Number analyzed (Participants) | 270 | 271 | 270
score on a scale | 22.8 (0.6) | 22.7 (0.6) | 24.9 (0.6)
Statistical Analysis 1: Comparison: Mobile+Group LAMP Mindfulness-Based Intervention vs Mobile LAMP Mindfulness-Based Intervention; Test type: Superiority; p = 0.886, Mixed Models Analysis; Linear mixed model adjusted for baseline values of PCL5, Pain Self-Efficacy, and design factors; Mean Difference (Final Values) = 0.1, 95% CI 2-sided [-1.6 to 1.9] — estimates were generated from multiple imputed data
Statistical Analysis 2: Comparison: Mobile+Group LAMP Mindfulness-Based Intervention vs Usual Care; Test type: Superiority; p = 0.017, Mixed Models Analysis; Linear mixed model adjusted for baseline values of PCL5, Pain Self-Efficacy, and design factors; Mean Difference (Final Values) = -2.0, 95% CI 2-sided [-3.7 to -0.4] — estimates were generated from multiple imputed data
Statistical Analysis 3: Comparison: Mobile LAMP Mindfulness-Based Intervention vs Usual Care; Test type: Superiority; p = 0.013, Mixed Models Analysis; Linear mixed model adjusted for baseline values of PCL5, Pain Self-Efficacy, and design factors; Mean Difference (Final Values) = -2.2, 95% CI 2-sided [-3.9 to -0.5] — estimates were generated from multiple imputed data

10. Secondary Outcome: Mean Global Improvement of Pain Score, Over the 12-month Follow-up Period
Description: Global impression of change scale from "much better" to "much worse". Minimum value: 1. Maximum value: 7. Higher scores indicate worse outcome. Change in the outcome measure operationalized as the weighted average of all of the time points during follow-up.
Time Frame: Weighted average over 10 weeks, 6 months, and 12 months.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Mobile+Group LAMP Mindfulness-Based Intervention | Mobile LAMP Mindfulness-Based Intervention | Usual Care
Number analyzed (Participants) | 270 | 271 | 270
units on a scale | 3.4 (0.1) | 3.3 (0.1) | 4.1 (0.1)
Statistical Analysis 1: Comparison: Mobile+Group LAMP Mindfulness-Based Intervention vs Mobile LAMP Mindfulness-Based Intervention; Test type: Superiority; p = 0.437, Mixed Models Analysis; Linear mixed model adjusted for baseline Pain Self-Efficacy, and design factors; Mean Difference (Final Values) = 0.1, 95% CI 2-sided [-0.1 to 0.3] — estimates were generated from multiple imputed data
Statistical Analysis 2: Comparison: Mobile+Group LAMP Mindfulness-Based Intervention vs Usual Care; Test type: Superiority; p < 0.001, Mixed Models Analysis; Linear mixed model adjusted for baseline Pain Self-Efficacy, and design factors; Mean Difference (Final Values) = -0.7, 95% CI 2-sided [-0.9 to -0.5] — estimates were generated from multiple imputed data
Statistical Analysis 3: Comparison: Mobile LAMP Mindfulness-Based Intervention vs Usual Care; Test type: Superiority; p < 0.001, Mixed Models Analysis; Linear mixed model adjusted for baseline Pain Self-Efficacy, and design factors; Mean Difference (Final Values) = -0.8, 95% CI 2-sided [-1.0 to -0.6] — estimates were generated from multiple imputed data

11. Secondary Outcome: BPI Interference Score Responder Analysis
Description: Change in Brief Pain Inventory (BPI) interference score over the 12-month follow-up period. Number with 30% improvement in BPI inference score. Change in the outcome measure operationalized as the weighted average of all of the time points during follow-up, adjusting for the baseline value prior to randomization.
Time Frame: Weighted average over 10 weeks, 6 months, and 12 months.
Measure: Count of Participants; unit: Participants
Arm/Group | Mobile+Group LAMP Mindfulness-Based Intervention | Mobile LAMP Mindfulness-Based Intervention | Usual Care
Number analyzed (Participants) | 270 | 271 | 270
Participants | 89 | 109 | 56
Statistical Analysis 1: Comparison: Mobile+Group LAMP Mindfulness-Based Intervention vs Mobile LAMP Mindfulness-Based Intervention; Test type: Superiority; Mixed Models Analysis — Used confidence interval to determine significance; Logistic mixed model adjusted for baseline values of BPI interference, Pain Self-Efficacy, and design factors; Mean Difference (Final Values) = -7.5, 95% CI 2-sided [-13.9 to -1.2] — estimates were generated from multiple imputed data
Statistical Analysis 2: Comparison: Mobile+Group LAMP Mindfulness-Based Intervention vs Usual Care; Test type: Superiority; Mixed Models Analysis — Used confidence interval to determine significance; Logistic mixed model adjusted for baseline values of BPI interference, Pain Self-Efficacy, and design factors; Mean Difference (Final Values) = 12.0, 95% CI 2-sided [6.4 to 17.6] — estimates were generated from multiple imputed data
Statistical Analysis 3: Comparison: Mobile LAMP Mindfulness-Based Intervention vs Usual Care; Test type: Superiority; Mixed Models Analysis — Used confidence interval to determine significance; Logistic mixed model adjusted for baseline values of BPI interference, Pain Self-Efficacy, and design factors; Mean Difference (Final Values) = 19.5, 95% CI 2-sided [13.6 to 25.4] — estimates were generated from multiple imputed data

ADVERSE EVENTS:
Time Frame: Adverse event data were collected for each participant from the time they completed the baseline survey through their final follow-up survey time period. This is equal to approximately 16 months for each participant depending when exactly they completed each survey.
Arm/Group | Mobile+Group LAMP Mindfulness-Based Intervention | Mobile LAMP Mindfulness-Based Intervention | Usual Care
All-Cause Mortality (participants affected / at risk) | 0/270 | 0/271 | 0/270
Serious Adverse Events (participants affected / at risk) | 0/270 | 0/271 | 0/270
Other Adverse Events (participants affected / at risk) | 0/270 | 0/271 | 0/270

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-04-08): https://cdn.clinicaltrials.gov/large-docs/58/NCT04526158/Prot_SAP_000.pdf